CLINICAL TRIAL: NCT03722199
Title: Effects of Flavanoids on Acute Peripheral Vascular Reactivity in Essential Hypertension, Type 2 Diabetes and Healthy Persons
Brief Title: Effects of Flavanoids in Essential Hypertension, Type 2 Diabetes and Healthy Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B670201835660
Record Dates: First submitted 2018-09-28; First posted 2018-10-26 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2020-08

CONDITIONS: Vascular Complications, Diabetic
Keywords: flavanols; diabetes type 2; essential hypertension; peripheral vascular function
MeSH Terms: conditions — Diabetic Angiopathies; Diabetes Mellitus, Type 2; Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The different capsules are separated into 2 boxes but both sorts of capsules have the same colour and size. They just have a different number marked on the white box. During the investigation day, the participant chooses an envelope marked with number 1 or number 2 leading to the decision of the box and thus the capsules they will get.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy persons (Experimental): In this interventional study the investigators ask the patient (healthy persons) to come twice. One time they get capsules (6 or 8) with real flavanols (subgroup of polyphenols, subgroup of phenolics, natural substances) and the other time they get capsules with a placebo
  Interventions: Dietary Supplement: flavanols (subgroup of polyphenols, subgroup of phenolics, natural substances); Other: Placebo
- Persons with essential hypertension (Experimental): In this interventional study the investigators ask the patient (persons with essential hypertension) to come twice. One time they get capsules (6 or 8) with real flavanols (subgroup of polyphenols, subgroup of phenolics, natural substances) and the other time they get capsules with a placebo
  Interventions: Dietary Supplement: flavanols (subgroup of polyphenols, subgroup of phenolics, natural substances); Other: Placebo
- Persons with type 2 diabetes (Experimental): In this interventional study the investigators ask the patient (persons with type 2 diabetes) to come twice. One time they get capsules (6 or 8) with real flavanols (subgroup of polyphenols, subgroup of phenolics, natural substances) and the other time they get capsules with a placebo
  Interventions: Dietary Supplement: flavanols (subgroup of polyphenols, subgroup of phenolics, natural substances); Other: Placebo

INTERVENTIONS:
Dietary Supplement: flavanols (subgroup of polyphenols, subgroup of phenolics, natural substances) — single intake of capsules with flavanols (subgroup of polyphenols, subgroup of phenolics, natural substances)
  Other Names: flavanoids
Other: Placebo — single intake of capsules with a placebo

SUMMARY:
Flavanols are natural substances who are frequently found in our nutrition. A lot of research has already been executed in the past to investigate what effects this flavanols could have in the human population. Based on these examinations, the investigators think and suggest that flavanols can have positive effects on the vascularly system, more specifically on the peripheral and cerebral blood vessels. The effects are only observed in a healthy populations, meanwhile patient populations like diabetes patients could really benefit from this. This is why the investigators will execute this study.

DETAILED DESCRIPTION:
The study population is divided into 3 main groups, namely healthy controls, patients with diabetes type 2 (defined by American Diabetes Association's (ADA)) and patients with essential hypertension (the latter group is again divided into 3 subgroups: use of betablockers, angiotensin-converting enzyme (ACE)-inhibitors, angiotensin-receptor blockers (ARBs). Each main goup will consist of minimal 20 subjects.

In this interventional study the investigators ask the patient to come twice. One time they get capsules with real flavanols and the other time they get capsules with a placebo. The study will be double blinded so nor the investigators, nor the patients now at which investigation they get the real flavanols or the placebo.

Before and after the intake of these capsules, a few measurements will take place. These measurements will be compared on the one hand with the second investigation day (inter-patients and intra-patient) and on the other hand with the pre-intake measurements (intra-patient).

The different examinations are a Flow-mediated dilatation (FMD) test, blood pressure analysis and an exercise test.

The investigator who performs the FMD-test, followed a course and needed to pass an examination.

The blood pressure measurements will be continuously for 20 minutes to avoid to much bias.

ELIGIBILITY:
Inclusion Criteria:

* men and woman, age 18 - 85 years old, diabetes type 2 and/or using 1 sort of blood pressure lowering medication (betablockers, calcium-antagonists, RAAS-inhibitors)

Exclusion Criteria:

* GENERAL: diabetes type 1, maturity-onset diabetes of youth (MODY), Latent Autoimmune Diabetes of the Adult (LADA), smokers, alcohol abuse, active cancer, chronic inflammatory disease
* MICROVASCULAR: retinopathy, diabetic/hypertensive nephropathy, peripheral sensoric neuropathy, autonomic neuropathy
* MACROVASCULAR: cardiovascular diseases, cerebrovascular diseases, active or chronic palindromic vasculitis
* MEDICATION with impact on endothelial function: NO-containing medication, phosphodiesterase Type 5 -inhibitors
* DISEASES who can affect the exercise test: chronic obstructive pulmonary disease (COPD) with Global Initiative for Chronic Obstructive Lung Disease (GLOD) -stages III and IV, Heart failure class 3 and 4, serious musculoskeletal diseases
* OTHER: pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
FMD -Flow mediated dilatation test | 20 minutes
  Flow mediated dilatation test

SECONDARY OUTCOMES:
blood pressure analysis | 25 minutes
  analysis of changes in systolic or diastolic blood pressure

OTHER OUTCOMES:
Near-infrared spectroscopy during exercise | 25 minutes
  analysis of changes in oxygenated blood during exercise
exercise test with hand held dynamometer | 25 minutes
  analysis of changes in maximal capacity

CONTACTS AND LOCATIONS:
Overall Officials: Samyah Shadid, Prof. Dr., Principal Investigator — Universal hospital of Ghent and university of Ghent
Locations (1):
- University of Ghent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tanghe A, Celie B, Shadid S, Rietzschel E, Op 't Roodt J, Reesink KD, Heyman E, Calders P. Acute Effects of Cocoa Flavanols on Blood Pressure and Peripheral Vascular Reactivity in Type 2 Diabetes Mellitus and Essential Hypertension: A Protocol for an Acute, Randomized, Double-Blinded, Placebo-Controlled Cross-Over Trial. Front Cardiovasc Med. 2021 Mar 15;8:602086. doi: 10.3389/fcvm.2021.602086. eCollection 2021. PMID 33791343